CLINICAL TRIAL: NCT02488408
Title: A Phase Ib/II Multicenter Open-label Study of BGB324 as a Single Agent and in Combination With Cytarabine or Decitabine in Patients With Acute Myeloid Leukemia or as a Single Agent in Patients With Myelodysplastic Syndrome
Brief Title: A Phase Ib/II Multicenter Open-label Study of Bemcentinib (BGB324) in Patients With AML or MDS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BerGenBio ASA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGBC003
Record Dates: First submitted 2015-04-23; First posted 2015-07-02 (Estimated); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: BGB324; bemcentinib
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — bemcentinib; Cytarabine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A (Experimental): Bemcentinib will be administered as monotherapy in participants with relapsed or refractory AML following previous treatment with cytotoxic chemotherapy (with or without hematopoietic stem cell transplantation) or a gene expression modulator, such as a demethylating agent.
  Interventions: Drug: Bemcentinib
- Part B1 (Experimental): Single agent bemcentinib will be administered to participants with AML who are unsuitable for intensive chemotherapy as a result of advanced age and/or existing co-morbidities.
  Interventions: Drug: Bemcentinib
- Part B2 (Experimental): Bemcentinib will be administered in combination with low dose cytarabine in participants with AML who are unsuitable for intensive chemotherapy as a result of advanced age or existing co-morbidities.
  Interventions: Drug: Bemcentinib; Drug: Cytarabine
- Part B3 (Experimental): Bemcentinib will be administered in combination with decitabine in participants with AML who are unsuitable for intensive chemotherapy as a result of advanced age or existing co-morbidities.
  Interventions: Drug: Bemcentinib; Drug: Decitabine
- Part B4 (Experimental): Bemcentinib will be administered as a monotherapy to participants with previously treated MDS (including high risk and intermediate with the exception of deletion 5q MDS).
  Interventions: Drug: Bemcentinib
- Part B5 (Experimental): Bemcentinib will be administered in combination with low dose cytarabine in participants with relapsed or refractory who have received at least one prior treatment for. Participants must be unsuitable for intensive chemotherapy as a results of advanced age or existing co-morbidities.
  Interventions: Drug: Bemcentinib; Drug: Cytarabine

INTERVENTIONS:
Drug: Bemcentinib
  Other Names: BGB324
Drug: Cytarabine
  Other Names: Ara-C
  Arms: Part B2; Part B5
Drug: Decitabine
  Other Names: Dacogen
  Arms: Part B3

SUMMARY:
A Phase Ib/II multicentre open label study of bemcentinib (BGB324) as a single agent in participants with Acute Myeloid Leukemia (AML) or Myelodysplastic syndrome (MDS) or in a combination with cytarabine or decitabine in AML participants.

Bemcentinib is a potent selective small molecule inhibitor of AXL a surface membrane protein kinase receptor which is overexpressed in up to half of AML cases.

DETAILED DESCRIPTION:
This study is a dose-escalation of bemcentinib (BGB324), a selective AXL kinase inhibitor, in participants with AML and MDS, followed by a cohort expansion study of bemcentinib either as a single agent in participants with AML or MDS, or in combination with cytarabine (cytosine arabinoside, Ara-C) or decitabine in participants with AML.

The study will run in Germany, Norway, Italy and the US and may enrol up to approximately 90 participants with AML or MDS.

The study consisted of a dose-escalation phase to determine the MTD (maximum tolerated dose) and/or recommended dose for Phase II (RP2D) of bemcentinib in participants with relapsed or refractory AML or MDS (Part A) followed by a cohort expansion phase in five disease-specific cohorts (Part B).

Bemcentinib was administered orally according to a daily schedule, with the first three doses of Cycle 1 serving as a 'loading' dose. Each 21-day (three week) period will constitute 1 cycle of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed written informed consent.
2. Histological, molecular or cytological confirmation of:

   1. Part A: Participants must have received previous treatment with cytotoxic chemotherapy (with or without hematopoietic stem cell transplantation) or a gene expression modulator, such as a demethylating agent. Participants suitable for intensive chemotherapy should be in second or subsequent relapse or be refractory to at least two induction regimens. If eligible they should have undergone hematopoietic stem cell transplantation. Participants receiving an allograft in first remission would be eligible at the time of relapse. Participants who are unsuitable for intensive chemotherapy as a result of advanced age or co-morbidities should have relapsed following at least one line of therapy or be refractory.
   2. Part B1: Participants with AML who are unsuitable for intensive chemotherapy as a result of advanced age or co-morbidities. Participants should have relapsed following at least one line of therapy or be refractory to such prior therapy. Participants should not have received standard dose intensive chemotherapy.
   3. Part B2: Participants with AML who are unsuitable for intensive chemotherapy as a result of advancing age or co-morbidities and who are suitable to receive treatment with cytarabine.
   4. Part B3: Participants with AML who are unsuitable for intensive chemotherapy as a result if advancing age or co-morbidities and who are suitable to receive treatment with decitabine.
   5. Part B4: Participants with MDS (with the exception of deletion 5q MDS) including intermediate and high-risk participants who must have received prior treatment for their disease. Prior treatment may include those participants who have received hypomethylating agents, decitabine or other approved treatments for MDS.
   6. Part B5: Participants with relapsed or refractory AML who are unsuitable for intensive chemotherapy as a result of advanced age or co-morbidities meeting the following criteria:

      * Must have received at least one prior treatment for AML Are suitable to receive treatment with "low-dose" cytarabine (LDAC). LDAC is defined as 20 mg cytarabine administered subcutaneously twice daily for 10 days every 28 days. The number of participants with refractory AML, defined as no hematological response to last AML treatment and/or participants who have received 2 or more prior treatments for AML, will be restricted to 1/3 of the sample size (i.e. no more than 6 evaluable participants).
3. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.
4. Age 18 years or older.
5. Female participants of childbearing potential must have a negative serum pregnancy test within 3 days prior to taking their first dose of bemcentinib. Male participants and female participants of reproductive potential must practice highly effective methods of contraception (such as hormonal implants, combined oral contraceptives, injectable contraceptives, intrauterine device with hormone spirals, total sexual abstinence, vasectomy) throughout the study and for >=3 months after the last dose of bemcentinib.

Female participants are considered NOT of childbearing potential if they have a history of surgical sterility or evidence of post-menopausal status defined as any of the following:

1. Natural menopause with last menses >1 year ago.
2. Radiation induced oophorectomy with last menses >1 year ago.
3. Chemotherapy induced menopause with last menses >1 year ago.

Exclusion Criteria:

1. Participants who have a matched donor and are candidates for allogeneic bone marrow transplantation.
2. Pregnant or lactating
3. History of the following cardiac conditions:

   * Congestive cardiac failure of >Class II severity according to the New York Heart Association (defined as symptomatic at less than ordinary levels of activity)
   * Ischemic cardiac event including myocardial infarction within 3 months prior to first dose. Participants with prior history or ECG evidence of old myocardial infarction should be discussed with the Sponsor to confirm eligibility.
   * Uncontrolled cardiac disease, including unstable angina, uncontrolled hypertension (i.e. sustained systolic BP >160 mmHg or diastolic BP >90 mmHg), or need to change medication within 6 weeks of provision of consent due to lack of BP control
   * History or presence of sustained bradycardia (<=55 beats per minute), left bundle branch block, cardiac pacemaker or ventricular arrhythmia.

   Note: Participants with supraventricular arrhythmia should be discussed with the Sponsor to confirm eligibility.
   * Family history of long QTc syndrome; personal history of long QTc syndrome or previous drug-induced QTc prolongation of at least Grade 3 (QTc >500 ms).
   * Presence of any factors that increase the risk for QTc prolongation, e.g. resistant or inadequately treated heart failure, presence of hypokalemia or hypomagnesemia not corrected by, or not responding to, replacement therapy or inadequately treated hypothyroidism as defined by the thyroid-stimulating hormone not within the expected range of the institution.
4. Abnormal left ventricular ejection fraction (less than the lower limit of normal for a participants of that age at the treating institution or <45%, whichever is lower).
5. Current treatment with any agent known to cause QT prolongation and have a risk for Torsades de Pointes which cannot be discontinued at least 5 half-lives or 2 weeks prior to the first dose of study treatment. Please see Appendix 3 for list of relevant medications.
6. Screening 12-lead ECG with a measurable QTcF >450 ms.
7. Ongoing infection requiring systemic treatment. participants who are on prophylactic antimicrobials or who have been afebrile for 48 hours following the initiation of antimicrobials are eligible.
8. Inadequate liver function as demonstrated by serum bilirubin >=1.5 times the upper limits of normal range (ULN) or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >=2.5 times the ULN (or >=5 times the ULN for AST or ALT in the presence of liver involvement by leukemia).
9. Inability to tolerate oral medication.
10. Existing gastrointestinal disease affecting drug absorption such as celiac disease or Crohn's disease.
11. Known lactose intolerance.
12. Requires vitamin K antagonists. Note: participants receiving low doses prescribed to maintain the patency of venous access devices may be included.
13. Treatment with any of the following H2 receptor antagonists, proton pump inhibitors or antacids within 3 days of administration of bemcentinib.
14. Treatment with any medication which is predominantly metabolized by CYP3A4 and has a narrow therapeutic index.
15. Previous bowel resection that would interfere with drug absorption.
16. Evidence of ongoing gastrointestinal graft versus host disease.
17. Hematopoietic stem cell transplantation within 6 months.
18. Impaired renal function as demonstrated by a creatinine clearance of <30 mL/min determined by Cockcroft-Gault formula.
19. Radiotherapy or chemotherapy within the 14 days prior to the first dose of bemcentinib being administered (other than hydroxyurea).
20. Receiving an investigational anti-cancer treatment concurrently or within 14 days or five half-lives (whichever is shorter) of either the parent drug or any known active metabolite prior to the start of bemcentinib.
21. Unresolved CTCAE >Grade 2 toxicity (other than stable toxicity) from previous anti-cancer therapy excluding alopecia.
22. Any evidence of severe or uncontrolled systemic conditions (e.g., severe hepatic impairment) or current unstable or uncompensated respiratory or cardiac conditions which makes it undesirable for the participants to participate in the study or which could jeopardize compliance with the protocol.
23. Active, uncontrolled central nervous system (CNS) disease including CNS leukemia.
24. Active infection with human immunodeficiency virus (HIV), hepatitis B or C viruses - screening for viral infections is not required for entry to this study.
25. Major surgery within 28 days prior to the start of bemcentinib - excluding skin biopsies and procedures for insertion of central venous access devices.
26. Hypersensitivity to cytarabine, decitabine or any of its excipients.
27. Prior exposure to Astellas ASP2215 (FLT3/AXL Inhibitor - Gilteritinib).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Loges, MD, Principal Investigator — Universitätsmedizin Mannheim, Universitätsklinikum Mannheim GmbH
Locations (12):
- United States (2):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
- Germany (5):
  - Medizinische Hochschule Hannover,Hämatologie, Hämostaseologie, Onkologie und Stammzelltransplantation,, Hanover, Carl-Neuberg-Str
  - University Medical Center Hamburg, Hamburg, Hamburg-Eppendorf
  - Frankfurt Medizinische Klinik II, Hämatologie/Onkologie, Haus 33, 2. OG, Frankfurt, Theodor-Stern-Kai
  - Studienzentrale der Hämatologie/Onkologie III, Medizinische Klinik, Mannheim
  - Universitätsklinikum Ulm, Ulm
- Italy (4):
  - Azienda Ospedaliera S Croce E Carle, Via Michele Coppino, Cuneo
  - Ospedale Policlinico San Martino, Genoa
  - Ospedale Lecce - 'V Fazzi' U. O. Ematologia - P. O. Vito Fazz Piazza Muratore, IV piano Polo Oncologico, Lecce
  - Azienda Ospedaliero-Universitaria di Parma, Parma
- University of Bergen Department of Clinical Science, Translational Hemato-Oncology group, Faculty of Medicine and Dentistry, Haukelands University Hospital, Bergen, Jonas Lies Vei, Norway

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification [text, tables, figures and appendices].
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Proposal should be directed to HYPERLINK "mailto:clinical@bergenbio.com" clinical@bergenbio.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Ben-Batalla I, Schultze A, Wroblewski M, Erdmann R, Heuser M, Waizenegger JS, Riecken K, Binder M, Schewe D, Sawall S, Witzke V, Cubas-Cordova M, Janning M, Wellbrock J, Fehse B, Hagel C, Krauter J, Ganser A, Lorens JB, Fiedler W, Carmeliet P, Pantel K, Bokemeyer C, Loges S. Axl, a prognostic and therapeutic target in acute myeloid leukemia mediates paracrine crosstalk of leukemia cells with bone marrow stroma. Blood. 2013 Oct 3;122(14):2443-52. doi: 10.1182/blood-2013-03-491431. Epub 2013 Aug 27. PMID 23982172
- [Background] Cheson BD, Bennett JM, Kopecky KJ, Buchner T, Willman CL, Estey EH, Schiffer CA, Doehner H, Tallman MS, Lister TA, Lo-Coco F, Willemze R, Biondi A, Hiddemann W, Larson RA, Lowenberg B, Sanz MA, Head DR, Ohno R, Bloomfield CD; International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. Revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. J Clin Oncol. 2003 Dec 15;21(24):4642-9. doi: 10.1200/JCO.2003.04.036. PMID 14673054
- [Background] Cheson BD, Greenberg PL, Bennett JM, Lowenberg B, Wijermans PW, Nimer SD, Pinto A, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Gore SD, Schiffer CA, Kantarjian H. Clinical application and proposal for modification of the International Working Group (IWG) response criteria in myelodysplasia. Blood. 2006 Jul 15;108(2):419-25. doi: 10.1182/blood-2005-10-4149. Epub 2006 Apr 11. PMID 16609072
- [Background] Dohner H, Estey E, Grimwade D, Amadori S, Appelbaum FR, Buchner T, Dombret H, Ebert BL, Fenaux P, Larson RA, Levine RL, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz M, Sierra J, Tallman MS, Tien HF, Wei AH, Lowenberg B, Bloomfield CD. Diagnosis and management of AML in adults: 2017 ELN recommendations from an international expert panel. Blood. 2017 Jan 26;129(4):424-447. doi: 10.1182/blood-2016-08-733196. Epub 2016 Nov 28. PMID 27895058
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Whitman SP, Kohlschmidt J, Maharry K, Volinia S, Mrozek K, Nicolet D, Schwind S, Becker H, Metzeler KH, Mendler JH, Eisfeld AK, Carroll AJ, Powell BL, Carter TH, Baer MR, Kolitz JE, Park IK, Stone RM, Caligiuri MA, Marcucci G, Bloomfield CD. GAS6 expression identifies high-risk adult AML patients: potential implications for therapy. Leukemia. 2014 Jun;28(6):1252-1258. doi: 10.1038/leu.2013.371. Epub 2013 Dec 11. PMID 24326683
- [Background] Linger RM, Keating AK, Earp HS, Graham DK. TAM receptor tyrosine kinases: biologic functions, signaling, and potential therapeutic targeting in human cancer. Adv Cancer Res. 2008;100:35-83. doi: 10.1016/S0065-230X(08)00002-X. PMID 18620092
- [Background] Linger RM, Keating AK, Earp HS, Graham DK. Taking aim at Mer and Axl receptor tyrosine kinases as novel therapeutic targets in solid tumors. Expert Opin Ther Targets. 2010 Oct;14(10):1073-90. doi: 10.1517/14728222.2010.515980. PMID 20809868
- [Background] Schmidt T, Ben-Batalla I, Schultze A, Loges S. Macrophage-tumor crosstalk: role of TAMR tyrosine kinase receptors and of their ligands. Cell Mol Life Sci. 2012 May;69(9):1391-414. doi: 10.1007/s00018-011-0863-7. Epub 2011 Nov 11. PMID 22076650
- [Background] Gjerdrum C, Tiron C, Hoiby T, Stefansson I, Haugen H, Sandal T, Collett K, Li S, McCormack E, Gjertsen BT, Micklem DR, Akslen LA, Glackin C, Lorens JB. Axl is an essential epithelial-to-mesenchymal transition-induced regulator of breast cancer metastasis and patient survival. Proc Natl Acad Sci U S A. 2010 Jan 19;107(3):1124-9. doi: 10.1073/pnas.0909333107. Epub 2009 Dec 28. PMID 20080645
- [Background] Korshunov VA. Axl-dependent signalling: a clinical update. Clin Sci (Lond). 2012 Apr;122(8):361-8. doi: 10.1042/CS20110411. PMID 22187964
- [Background] Zhang Z, Lee JC, Lin L, Olivas V, Au V, LaFramboise T, Abdel-Rahman M, Wang X, Levine AD, Rho JK, Choi YJ, Choi CM, Kim SW, Jang SJ, Park YS, Kim WS, Lee DH, Lee JS, Miller VA, Arcila M, Ladanyi M, Moonsamy P, Sawyers C, Boggon TJ, Ma PC, Costa C, Taron M, Rosell R, Halmos B, Bivona TG. Activation of the AXL kinase causes resistance to EGFR-targeted therapy in lung cancer. Nat Genet. 2012 Jul 1;44(8):852-60. doi: 10.1038/ng.2330. PMID 22751098
- [Background] Byers LA, Diao L, Wang J, Saintigny P, Girard L, Peyton M, Shen L, Fan Y, Giri U, Tumula PK, Nilsson MB, Gudikote J, Tran H, Cardnell RJ, Bearss DJ, Warner SL, Foulks JM, Kanner SB, Gandhi V, Krett N, Rosen ST, Kim ES, Herbst RS, Blumenschein GR, Lee JJ, Lippman SM, Ang KK, Mills GB, Hong WK, Weinstein JN, Wistuba II, Coombes KR, Minna JD, Heymach JV. An epithelial-mesenchymal transition gene signature predicts resistance to EGFR and PI3K inhibitors and identifies Axl as a therapeutic target for overcoming EGFR inhibitor resistance. Clin Cancer Res. 2013 Jan 1;19(1):279-90. doi: 10.1158/1078-0432.CCR-12-1558. Epub 2012 Oct 22. PMID 23091115
- [Background] Safaric Tepes P, Pal D, Lindsted T, Ibarra I, Lujambio A, Jimenez Sabinina V, Senturk S, Miller M, Korimerla N, Huang J, Glassman L, Lee P, Zeltsman D, Hyman K, Esposito M, Hannon GJ, Sordella R. An epigenetic switch regulates the ontogeny of AXL-positive/EGFR-TKi-resistant cells by modulating miR-335 expression. Elife. 2021 Jul 13;10:e66109. doi: 10.7554/eLife.66109. PMID 34254585
- [Background] Meel MH, de Gooijer MC, Metselaar DS, Sewing ACP, Zwaan K, Waranecki P, Breur M, Buil LCM, Lagerweij T, Wedekind LE, Twisk JWR, Koster J, Hashizume R, Raabe EH, Montero Carcaboso A, Bugiani M, Phoenix TN, van Tellingen O, van Vuurden DG, Kaspers GJL, Hulleman E. Combined Therapy of AXL and HDAC Inhibition Reverses Mesenchymal Transition in Diffuse Intrinsic Pontine Glioma. Clin Cancer Res. 2020 Jul 1;26(13):3319-3332. doi: 10.1158/1078-0432.CCR-19-3538. Epub 2020 Mar 12. PMID 32165429
- [Derived] Loges S, Heuser M, Chromik J, Sutamtewagul G, Kapp-Schwoerer S, Crugnola M, Di Renzo N, Lemoli R, Mattei D, Fiedler W, Alvarado-Valero Y, Ben-Batalla I, Waizenegger J, Rieckmann LM, Janning M, Collienne M, Imbusch CD, Beumer N, Micklem D, H Nilsson L, Madeleine N, McCracken N, Oliva C, Gorcea-Carson C, Gjertsen BT. Bemcentinib as monotherapy and in combination with low-dose cytarabine in acute myeloid leukemia patients unfit for intensive chemotherapy: a phase 1b/2a trial. Nat Commun. 2025 Mar 23;16(1):2846. doi: 10.1038/s41467-025-58179-6. PMID 40122885
- See also: Please see BerGenBio's website for more information. — http://www.bergenbio.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 122 participants were enrolled to the study and received study treatment.
Groups:
- Part A: Bemcentinib 400/100 Milligram (mg): Participants with relapsed or refractory acute myeloid leukemia (AML) who received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 100 mg thereafter. Each cycle was of 21 days. Maximum exposure was of 568 days.
- Part A: Bemcentinib 600/200 mg: Participants with relapsed or refractory AML initially received loading dose of bemcentinib 600 mg on Days 1 and 2. However, following the report of DLTs, subjects received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Each cycle was of 21 days. Maximum exposure was of 126 days. Hence, some participants received 600 mg and some received 400 mg of bemcentinib as loading dose.
- Part A: Bemcentinib 900/300 mg: Participants with relapsed or refractory AML initially received loading dose of bemcentinib 900 mg on Days 1 and 2. However, following the report of DLTs, participants received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Each cycle was of 21 days. Maximum exposure was of 122 days. Hence, some participants received 900 mg and some received 400 mg of bemcentinib as loading dose.
- Part A: Bemcentinib 200/100 mg: Participants with relapsed or refractory AML received daily loading dose of bemcentinib 200 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 100 mg thereafter. Each cycle was of 21 days. Maximum exposure was of 68 days.
- Part A: Bemcentinib 400/200 mg: Participants with relapsed or refractory AML who received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Each cycle was of 21 days. Maximum exposure was of 717 days.
- Part B1: Bemcentinib 400/200 mg: Participants with AML who are unsuitable for intensive chemotherapy, as a result of advanced age and/or existing co-morbidities and should have relapsed following at least one line of therapy or be refractory to such prior therapy received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Each cycle was of 21 days. Maximum exposure was of 602 days.
- Part B2: Bemcentinib 400/200 mg + Cytarabine: Participants with AML who are unsuitable for intensive chemotherapy, due to advanced age and/or existing co-morbidities, received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Each cycle was of 21 days. Maximum exposure to treatment was of 1424 days. In combination to this, participants received cytarabine subcutaneously according to standard practice (20 mg/m2 twice daily for 10 days followed by a rest period of <1 month according to persisting myelosuppression).
- Part B3: Bemcentinib 400/200 mg + Decitabine: Participants with AML who are unsuitable for intensive chemotherapy, due to advanced age and/or existing co-morbidities, received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Each cycle was of 21 days. Maximum exposure to treatment was of 393 days. In combination to this, participants received decitabine (up to a maximum dose of 20 mg/m2 body surface area by intravenous infusion over one hour, repeated daily for five consecutive days [i.e., a total of five doses per treatment cycle]).
- Part B4: Bemcentinib 400/200 mg: Participants with previously treated myelodysplastic syndrome (MDS) (with the exception of deletion 5q MDS) including intermediate (int-2) or high-risk MDS and who received prior treatment for the same. Prior treatment included participants who received hypomethylating agents, decitabine or other approved treatments for MDS. Participants received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Each cycle was of 21 days. Maximum exposure to treatment was of 449 days.
- Part B5: Bemcentinib 400/200 mg + Cytarabine: Participants with relapsed or refractory AML who are unsuitable for intensive chemotherapy, due to advanced age and/or existing co-morbidities who must have received at least one prior treatment for AML, received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Each cycle was of 21 days. Maximum exposure to treatment was of 462 days. In combination to this, participants received low dose cytarabine subcutaneously according to standard practice (dose of 20 mg subcutaneously twice daily for 10 days every 28 days).
Period: Part A
Arm/Group | Part A: Bemcentinib 400/100 Milligram (mg) | Part A: Bemcentinib 600/200 mg | Part A: Bemcentinib 900/300 mg | Part A: Bemcentinib 200/100 mg | Part A: Bemcentinib 400/200 mg | Part B1: Bemcentinib 400/200 mg | Part B2: Bemcentinib 400/200 mg + Cytarabine | Part B3: Bemcentinib 400/200 mg + Decitabine | Part B4: Bemcentinib 400/200 mg | Part B5: Bemcentinib 400/200 mg + Cytarabine
Started | 6 | 14 | 5 | 4 | 7 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 14 | 5 | 4 | 7 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 5 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 2 | 8 | 2 | 3 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Initiation of Alternative Cancer Therapy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator Decision | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Part A: Bemcentinib 400/100 Milligram (mg) | Part A: Bemcentinib 600/200 mg | Part A: Bemcentinib 900/300 mg | Part A: Bemcentinib 200/100 mg | Part A: Bemcentinib 400/200 mg | Part B1: Bemcentinib 400/200 mg | Part B2: Bemcentinib 400/200 mg + Cytarabine | Part B3: Bemcentinib 400/200 mg + Decitabine | Part B4: Bemcentinib 400/200 mg | Part B5: Bemcentinib 400/200 mg + Cytarabine
Started | 0 | 0 | 0 | 0 | 0 | 14 (Part B of the study had separate participants enrolled.) | 16 (Part B of the study had separate participants enrolled.) | 18 (Part B of the study had separate participants enrolled.) | 18 (Part B of the study had separate participants enrolled.) | 20 (Part B of the study had separate participants enrolled.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 14 | 16 | 18 | 18 | 20
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 7 | 2 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 2 | 2
Not completed — Death due to Disease Progression | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 1
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 6 | 9 | 7 | 9 | 11
Not completed — Initiation of Alternative Cancer Therapy | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 3
Not completed — Investigator Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAS) included all enrolled participants who received at least one dose of bemcentinib.
Groups:
- Part A: Bemcentinib 400/100 mg: Participants with relapsed or refractory AML who received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 100 mg thereafter. Each cycle was of 21 days. Maximum exposure was of 568 days.
- Part B1: Bemcentinib 400/200 mg, AML 400/200 mg Single Agent: Participants with AML who are unsuitable for intensive chemotherapy, as a result of advanced age and/or existing co-morbidities and should have relapsed following at least one line of therapy or be refractory to such prior therapy received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Each cycle was of 21 days. Maximum exposure was of 602 days.
- Part B2: Bemcentinib 400/200 mg + Cytarabine, AML: Participants with AML who are unsuitable for intensive chemotherapy, due to advanced age and/or existing co-morbidities, received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Each cycle was of 21 days. Maximum exposure to treatment was of 1424 days. In combination to this, participants received cytarabine subcutaneously according to standard practice (20 mg/m2 twice daily for 10 days followed by a rest period of <1 month according to persisting myelosuppression).
- Part B3: BGB324 400/200 mg + Decitabine, AML: Participants with AML who are unsuitable for intensive chemotherapy, due to advanced age and/or existing co-morbidities, received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Each cycle was of 21 days. Maximum exposure to treatment was of 393 days. In combination to this, participants received decitabine (up to a maximum dose of 20 mg/m2 body surface area by intravenous infusion over one hour, repeated daily for five consecutive days [i.e., a total of five doses per treatment cycle]).
- Part B4: BGB324 400/200 mg, MDS: Participants with previously treated MDS (with the exception of deletion 5q MDS) including intermediate (int-2) or high-risk MDS and who received prior treatment for the same. Prior treatment included participants who received hypomethylating agents, decitabine or other approved treatments for MDS. Participants received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Each cycle was of 21 days. Maximum exposure to treatment was of 449 days.
- Part B5: BGB324 400/200 mg + Cytarabine, AML: Participants with relapsed or refractory AML who are unsuitable for intensive chemotherapy, due to advanced age and/or existing co-morbidities who must have received at least one prior treatment for AML, received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Each cycle was of 21 days. Maximum exposure to treatment was of 462 days. In combination to this, participants received low dose cytarabine subcutaneously according to standard practice (dose of 20 mg subcutaneously twice daily for 10 days every 28 days).
- Total: Total of all reporting groups
Arm/Group | Part A: Bemcentinib 400/100 mg | Part A: Bemcentinib 600/200 mg | Part A: Bemcentinib 900/300 mg | Part A: Bemcentinib 200/100 mg | Part A: Bemcentinib 400/200 mg | Part B1: Bemcentinib 400/200 mg, AML 400/200 mg Single Agent | Part B2: Bemcentinib 400/200 mg + Cytarabine, AML | Part B3: BGB324 400/200 mg + Decitabine, AML | Part B4: BGB324 400/200 mg, MDS | Part B5: BGB324 400/200 mg + Cytarabine, AML | Total
Number analyzed (Participants) | 6 | 14 | 5 | 4 | 7 | 14 | 16 | 18 | 18 | 20 | 122
Age, Customized [Count of Participants; unit: Participants]
  <75 years | 3 | 8 | 3 | 2 | 2 | 6 | 5 | 3 | 9 | 7 | 48
  >= 75 years | 3 | 6 | 2 | 2 | 5 | 8 | 11 | 15 | 9 | 13 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 0 | 4 | 4 | 4 | 6 | 8 | 8 | 44
  Male | 3 | 11 | 1 | 4 | 3 | 10 | 12 | 12 | 10 | 12 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 6 | 14 | 5 | 4 | 7 | 14 | 15 | 18 | 17 | 20 | 120
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  White | 5 | 14 | 5 | 4 | 7 | 14 | 16 | 17 | 17 | 20 | 119
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part A: Maximum Tolerated Dose (MTD) of Bemcentinib (BGB324)
Description: If 1 participant in a cohort experienced a dose limiting toxicity (DLT) during Cycle 1, the cohort was expanded to 6 participants. If 2 of 3 or 2 of 6 participants in a cohort experience DLT no further dose escalation took place and the dose below was nominated as the MTD. DLT was assessed during the first 3 weeks of treatment (Cycle 1) with bemcentinib. DLT was defined as according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) [NCI CTCAE] version 4, considered unrelated to leukemia progression or intercurrent illness.
Time Frame: Cycle 1 (21 days)
Population: The safety analysis population in Part A included all enrolled participants who received at least one dose of bemcentinib in Part A.
Measure: Number; unit: mg
Groups:
- Part A: Bemcentinib: Participants who received bemcentinib in Part A of the study.
Arm/Group | Part A: Bemcentinib
Number analyzed (Participants) | 36
mg
  Loading dose for 3 days | 600
  Maintenance dose | 200

2. Primary Outcome: Part B: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant administered a pharmaceutical product and which did not necessarily had a causal relationship with the product. A TEAE was defined as an AE that started or worsened after the first dose of the study intervention until 28 days after the last dose.
Time Frame: Up to 28 days after last dose (up to 1452 days; maximum treatment exposure duration 1424 days)
Population: The safety analysis population in Part B included all enrolled participants who received at least one dose of bemcentinib in Part B.
Measure: Count of Participants; unit: Participants
Groups:
- Part B1: Bemcentinib 400/200 mg, AML: Participants with AML who are unsuitable for intensive chemotherapy, as a result of advanced age and/or existing co-morbidities and should have relapsed following at least one line of therapy or be refractory to such prior therapy received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Each cycle was of 21 days. Maximum exposure was of 602 days.
- Part B3: Bemcentinib 400/200 mg + Decitabine, AML: Participants with AML who are unsuitable for intensive chemotherapy, due to advanced age and/or existing co-morbidities, received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Each cycle was of 21 days. Maximum exposure to treatment was of 393 days. In combination to this, participants received decitabine (up to a maximum dose of 20 mg/m2 body surface area by intravenous infusion over one hour, repeated daily for five consecutive days [i.e., a total of five doses per treatment cycle]).
- Part B4: Bemcentinib 400/200 mg, MDS: Participants with previously treated MDS (with the exception of deletion 5q MDS) including intermediate (int-2) or high-risk MDS and who received prior treatment for the same. Prior treatment included participants who received hypomethylating agents, decitabine or other approved treatments for MDS. Participants received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Each cycle was of 21 days. Maximum exposure to treatment was of 449 days.
- Part B5: Bemcentinib 400/200 mg + Cytarabine, AML: Participants with relapsed or refractory AML who are unsuitable for intensive chemotherapy, due to advanced age and/or existing co-morbidities who must have received at least one prior treatment for AML, received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Each cycle was of 21 days. Maximum exposure to treatment was of 462 days. In combination to this, participants received low dose cytarabine subcutaneously according to standard practice (dose of 20 mg subcutaneously twice daily for 10 days every 28 days).
Arm/Group | Part B1: Bemcentinib 400/200 mg, AML | Part B2: Bemcentinib 400/200 mg + Cytarabine, AML | Part B3: Bemcentinib 400/200 mg + Decitabine, AML | Part B4: Bemcentinib 400/200 mg, MDS | Part B5: Bemcentinib 400/200 mg + Cytarabine, AML
Number analyzed (Participants) | 14 | 16 | 18 | 18 | 20
Participants | 14 | 16 | 18 | 18 | 20

3. Primary Outcome: Part B: Number of Participants With Notable Trends in Physical Examination, Vital Signs, Clinical Laboratory Test and Electrocardiogram (ECG) Values
Description: Number of participants with notable trends in physical examinations (including weight), vital signs (blood pressure [BP], heart rate [HR]), clinical laboratory test (including clinical chemistry, hematology and urinalysis), and ECG values over the time were reported in this outcome measure. Notable trends were defined as observations which were outside the normal range for these mentioned parameters as specified by the sponsor.
Time Frame: Baseline to end of the study (Part B: Maximum exposure duration was 1424 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part B1: Bemcentinib 400/200 mg, AML | Part B2: Bemcentinib 400/200 mg + Cytarabine, AML | Part B3: Bemcentinib 400/200 mg + Decitabine, AML | Part B4: Bemcentinib 400/200 mg, MDS | Part B5: Bemcentinib 400/200 mg + Cytarabine, AML
Number analyzed (Participants) | 14 | 16 | 18 | 18 | 20
Participants | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Part A: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: as for outcome 2
Time Frame: Up to 28 days after last dose (up to 745 days, maximum exposure duration 717 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Bemcentinib 400/100 mg | Part A: Bemcentinib 600/200 mg | Part A: Bemcentinib 900/300 mg | Part A: Bemcentinib 200/100 mg | Part A: Bemcentinib 400/200 mg
Number analyzed (Participants) | 6 | 14 | 5 | 4 | 7
Participants | 5 | 14 | 5 | 4 | 7

5. Secondary Outcome: Part A: Number of Participants With Notable Trends in Physical Examination, Vital Signs, Clinical Laboratory Test and Electrocardiogram (ECG) Values
Description: Number of participants with notable trends in physical examinations (including weight), vital signs (blood pressure [BP], heart rate [HR]), clinical laboratory test (including clinical chemistry, hematology and urinalysis), and ECG values over the time were reported as per investigator observation. Notable trends meant observations that were outside normal range as specified by sponsor.
Time Frame: Baseline to end of the study (Part A: Maximum exposure duration was 717 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Bemcentinib 400/100 mg | Part A: Bemcentinib 600/200 mg | Part A: Bemcentinib 900/300 mg | Part A: Bemcentinib 200/100 mg | Part A: Bemcentinib 400/200 mg
Number analyzed (Participants) | 6 | 14 | 5 | 4 | 7
Participants | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Part A and B: Percentage of Participants With Objective Response (OR) as Per International Working Group Response Criteria
Description: AML: complete remission (CR): Bone marrow (BM) <5% & no myeloblasts with Auer rods; absolute neutrophil count(ANC) >=1.0*10^9/L or >=1000/μL; platelet count (PC) >=100*10^9/L or >=100000/μL:CR with incomplete hematologic recovery(CRi): BM <5% and no myeloblasts with Auer rods; ANC <1.0*10^9/L or <1000/μL; PC <100*10^9/L or <100000/μL, CR with partial hematologic recovery (CRh): CR but ANC > 0.5 × 10^9/L and PC > 50 × 10^9/L; partial remission (PR): all CR hematologic criteria but decrease of myeloblasts to 5% to 25% and of pretreatment myeloblasts % by >= 50%; MDS: CR: BM <=5% myeloblasts, normal maturation of all cell lines, no evidence for dysplasia, Hb >=11 g/dL;PC >=100*10^9/L or 100000/μL; ANC >=1.5*10^9/L or 1500/μL; PB 0%; marrow CR: <=5% myeloblasts & decrease by >=50% over pretreatment value; CRh =CR with ANC > 0.5*10^9/L and PC > 50*10^9/L; PR: decrease of myeloblasts to 5% to 25% & decrease of pretreatment myeloblast by >= 50%; all hematologic criteria of CR.
Time Frame: Day 1 of dosing up to end of the study (for Part A: maximum exposure duration 717 days, and for Part B: maximum exposure duration 1424 days)
Population: Efficacy population included all participants from safety analysis population that met key eligibility criteria, have assessable disease at baseline and had at least 1 post-baseline response assessment; had received >1 dose of bemcentinib (and combination agent in Part B2, B3 and B5).
Measure: Number; unit: Percentage of participants
Groups:
- Part A: BGB324 200/100 mg: Participants with relapsed or refractory AML received daily loading dose of bemcentinib 200 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 100 mg thereafter. Each cycle was of 21 days. Maximum exposure was of 68 days.
Arm/Group | Part A: Bemcentinib 400/100 mg | Part A: Bemcentinib 600/200 mg | Part A: Bemcentinib 900/300 mg | Part A: BGB324 200/100 mg | Part A: Bemcentinib 400/200 mg | Part B1: Bemcentinib 400/200 mg, AML | Part B2: Bemcentinib 400/200 mg + Cytarabine, AML | Part B3: Bemcentinib 400/200 mg + Decitabine, AML | Part B4: Bemcentinib 400/200 mg, MDs | Part B5: Bemcentinib 400/200 mg + Cytarabine, AML
Number analyzed (Participants) | 3 | 10 | 4 | 4 | 6 | 11 | 14 | 13 | 16 | 18
Percentage of participants | 33.3 | 20.0 | 0 | 0 | 33.3 | 18.2 | 35.7 | 0 | 18.8 | 16.7

7. Secondary Outcome: Part A and B: Percentage of Participants With Stable Disease (SD) as Per International Working Group Response Criteria
Description: AML: SD= unchanged disease for at least 3 treatment cycles; MDS: SD = failure to achieve at least PR but no evidence of PD for at least 3 treatment cycles. AML: Absence of CR, Cri or PR and criteria for PD not met. MDS: PR = all CR criteria met if abnormal before treatment except for, myeloblasts decrease by 50% or more over pretreatment value but still >5%, or less advanced French-American-British (FAB) or International Prognostic Scoring System (IPPS) category compared to pretreatment value; hematologic improvement; absolute values must last at least 6 weeks. MDS: PD = for participants with <5% myeloblasts: a 50% or more increase in myeloblasts to more than 5% myeloblasts, for participants with 5% to 10% myeloblasts: a 50% or more increase to more than 10% myeloblasts, for participants with 10% to 20% myeloblasts: a 50% or more increase to more than 20% myeloblasts, for participants with 20% to 30% myeloblasts: a 50% or more increase to more than 30% myeloblasts.
Time Frame: as for outcome 6
Population: Efficacy population analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Bemcentinib 400/100 mg | Part A: Bemcentinib 600/200 mg | Part A: Bemcentinib 900/300 mg | Part A: Bemcentinib 200/100 mg | Part A: Bemcentinib 400/200 mg | Part B1: Bemcentinib 400/200 mg, AML | Part B2: Bemcentinib 400/200 mg + Cytarabine, AML | Part B3: Bemcentinib 400/200 mg + Decitabine, AML | Part B4: Bemcentinib 400/200 mg, MDS | Part B5: Bemcentinib 400/200 mg + Cytarabine, AML
Number analyzed (Participants) | 3 | 10 | 4 | 4 | 6 | 11 | 14 | 13 | 16 | 18
Percentage of participants | 0 | 0 | 25.0 | 25.0 | 0 | 27.3 | 14.3 | 30.8 | 37.5 | 0

8. Secondary Outcome: Part A and B: Disease Control Rate (DCR) as Per International Working Group Response Criteria
Description: AML and MDS: DCR= percentage of participants with OR and SD. AML: OR= CR, CRi, CRp, CRh and PR. MDS: OR= CR, PR, MR, PMR. AML: SD = unchanged disease for at least 3 treatment cycles; MDS: SD = failure to achieve at least PR but not evidence of PD for at least 3 treatment cycles.
Time Frame: as for outcome 6
Population: Efficacy population analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Bemcentinib 400/100 mg | Part A: Bemcentinib 600/200 mg | Part A: Bemcentinib 900/300 mg | Part A: Bemcentinib 200/100 mg | Part A: Bemcentinib 400/200 mg | Part B1: Bemcentinib 400/200 mg, AML | Part B2: Bemcentinib 400/200 mg + Cytarabine, AML | Part B3: Bemcentinib 400/200 mg + Decitabine, AML | Part B4: Bemcentinib 400/200 mg, MDS | Part B5: Bemcentinib 400/200 mg + Cytarabine, AML
Number analyzed (Participants) | 3 | 10 | 4 | 4 | 6 | 11 | 14 | 13 | 16 | 18
Percentage of participants | 33.3 | 20.0 | 25.0 | 25.0 | 33.3 | 45.5 | 50.0 | 30.8 | 56.3 | 16.7

9. Secondary Outcome: Part B: Relapse Free Survival (RFS)
Description: RFS: defined as the months from the date of response until the date of relapse as confirmed by blast counts assessment (date of the disease progression was used since disease progression is based in blast count assessment).
Time Frame: Day 1 of dosing up to end of the study (Part B: maximum exposure duration 1424 days)
Population: Efficacy population analyzed. "Overall Number of Participants Analyzed": Participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Part B1: Bemcentinib 400/200 mg, AML | Part B2: Bemcentinib 400/200 mg + Cytarabine, AML | Part B3: Bemcentinib 400/200 mg + Decitabine, AML | Part B4: Bemcentinib 400/200 mg, MDS | Part B5: Bemcentinib 400/200 mg + Cytarabine, AML
Number analyzed (Participants) | 2 | 5 | 0 | 3 | 3
Months | 6.61 [2.2 to 11.0] | 17.25 [2.3 to 44.7] |  | 3.08 [2.1 to 6.5] | 3.05 [2.6 to 12.9]

10. Secondary Outcome: Part B: Event Free Survival (EFS)
Description: Event was defined as death or progression. Duration of EFS was calculated as (days)= Date of onset of Event, subject death or censoring - Date of first intake of study treatment (Bemcentinib ) + 1. EFS data reported below is in months.
Time Frame: Day 1 of dosing up to end of the study (Part B: maximum exposure duration 1424 days)
Population: Efficacy population analyzed.
Measure: Median (Full Range); unit: Months
Arm/Group | Part B1: Bemcentinib 400/200 mg, AML | Part B2: Bemcentinib 400/200 mg + Cytarabine, AML | Part B3: Bemcentinib 400/200 mg + Decitabine, AML | Part B4: Bemcentinib 400/200 mg, MDS | Part B5: Bemcentinib 400/200 mg + Cytarabine, AML
Number analyzed (Participants) | 11 | 14 | 13 | 16 | 18
Months | 2.69 [0.7 to 18.7] | 3.75 [0.7 to 46.7] | 4.13 [1.4 to 12.5] | 4.18 [0.7 to 28.1] | 2.33 [0.7 to 21.3]

11. Secondary Outcome: Part B: Overall Survival (OS)
Description: OS was defined as the months from the first day of treatment until date of death for any cause. Participants who were alive at the time of the final analysis were censored at the date the participants were known to be alive.
Time Frame: Day 1 of dosing up to end of the study (Part B: maximum exposure duration 1424 days)
Population: Efficacy population analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B1: Bemcentinib 400/200 mg, AML | Part B2: Bemcentinib 400/200 mg + Cytarabine, AML | Part B3: Bemcentinib 400/200 mg + Decitabine, AML | Part B4: Bemcentinib 400/200 mg, MDS | Part B5: Bemcentinib 400/200 mg + Cytarabine, AML
Number analyzed (Participants) | 11 | 14 | 13 | 16 | 18
Months | 18.0 [2.7 to 20.5] | 11.1 [3.9 to 24.7] | 6.4 [3.3 to 11.6] | 9.2 [4.6 to 34.0] | 8.0 [2.5 to 21.3]

12. Secondary Outcome: Part A and Part B: Pharmacokinetics (PK) Parameter: Area Under The Curve (0-tau) at Steady State (AUCss) for Bemcentinib
Description: Predicted AUCss = area under the curve PK -time profile during 24 hours at steady state.
Time Frame: Predose, 2, 4, 6 hours post dose on Day 1;predose and 6hours post dose on Day2, predose, 2,4,6,8 hours post dose on Day 3 and predose on Day 4 of Cycle 1; Predose collected on Day1 of each cycle up to and including Cycle 15 and at end of the study (EOS)
Population: PK analysis population=participants who had 1 dose of bemcentinib & evaluable PK data available. Part A arms combined based on maintenance dose. Part B was not combined as combinations were different or were for different indications; time to attaining steady state affected by magnitude of loading dose, exposure at steady state would only be determined by level of daily maintenance dose. As pre-specified in analysis plan, data for arms that received same maintenance dose were reported combined.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Groups:
- Part A: Bemcentinib 400/100 mg + 200/100 mg: Participants received daily maintenance dose of 100 mg after Day 3 of Cycle 1 (21 days).
- Part A: Bemcentinib 600/200 mg + 400/200 mg: Participants received daily maintenance dose of 200 mg after Day 3 of Cycle 1 (21 days).
- Part A: Bemcentinib 900/300 mg: Participants received maintenance dose of 300 mg after Day 3 of Cycle 1 (21 days).
Arm/Group | Part A: Bemcentinib 400/100 mg + 200/100 mg | Part A: Bemcentinib 600/200 mg + 400/200 mg | Part A: Bemcentinib 900/300 mg | Part B1: Bemcentinib 400/200 mg, AML | Part B2: Bemcentinib 400/200 mg + Cytarabine, AML | Part B3: Bemcentinib 400/200 mg + Decitabine, AML | Part B4: Bemcentinib 400/200 mg, MDS | Part B5: Bemcentinib 400/200 mg + Cytarabine, AML
Number analyzed (Participants) | 10 | 21 | 5 | 14 | 15 | 17 | 17 | 20
nanogram*hour per milliliter (ng*h/mL) | 3310 (2630) | 3810 (2860) | 9390 (4720) | 4910 (2560) | 4650 (3260) | 5320 (2380) | 3510 (2010) | 5090 (2910)

13. Secondary Outcome: Part A and B: Pharmacokinetics Parameter: Maximum Observed Plasma Concentration (Cmax) for Bemcentinib
Description: Observed maximum predicted PK concentration (Cmax) during 24 hours at steady state (Cmax, ss).
Time Frame: Pre-dose 2, 4, 6 on Day 1; predose and 6 hours post dose on Day 2; predose, 2, 4, 6 and 8 hours post dose on Day 3 and predose on Day 4 of Cycle 1; Predose collected on Day 1 of each cycle up to and including Cycle 15 and at EOS
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A: Bemcentinib 400/100 mg + 200/100 mg | Part A: Bemcentinib 600/200 mg + 400/200 mg | Part A: Bemcentinib 900/300 mg | Part B1: Bemcentinib 400/200 mg, AML | Part B2: Bemcentinib 400/200 mg + Cytarabine, AML | Part B3: Bemcentinib 400/200 mg + Decitabine, AML | Part B4: Bemcentinib 400/200 mg, MDS | Part B5: Bemcentinib 400/200 mg + Cytarabine, AML
Number analyzed (Participants) | 10 | 21 | 5 | 14 | 15 | 17 | 17 | 20
nanogram per milliliter (ng/mL) | 140 (110) | 162 (121) | 398 (200) | 210 (108) | 198 (137) | 228 (101) | 150 (84.7) | 219 (123)

14. Secondary Outcome: Part A and B: Pharmacokinetics Parameter: t1/2 for Bemcentinib
Description: Median half-life (t1/2) at steady state.
Time Frame: as for outcome 13
Population: as for outcome 12
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: Bemcentinib 400/100 mg + 200/100 mg | Part A: Bemcentinib 600/200 mg + 400/200 mg | Part A: Bemcentinib 900/300 mg | Part B1: Bemcentinib 400/200 mg, AML | Part B2: Bemcentinib 400/200 mg + Cytarabine, AML | Part B3: Bemcentinib 400/200 mg + Decitabine, AML | Part B4: Bemcentinib 400/200 mg, MDS | Part B5: Bemcentinib 400/200 mg + Cytarabine, AML
Number analyzed (Participants) | 10 | 21 | 5 | 14 | 15 | 17 | 17 | 20
hours | 159 [67.5 to 608] | 124 [31.4 to 405] | 156 [87.3 to 384] | 157 [45.2 to 455] | 126 [58.2 to 362] | 155 [68.8 to 516] | 116 [43.6 to 507] | 112 [49.8 to 237]

ADVERSE EVENTS:
Time Frame: Up to 28 days after last dose (for Part A: up to 745 days, maximum exposure duration 717 days, and for Part B: up to 1452 days, maximum exposure duration1424 days)
Description: Adverse events were collected based on intervention (dose group) participants were initially assigned to receive, irrespective of loading or maintenance dose de-escalation if it occurred. SAS analyzed by dose group or combination in Part B.
Groups:
- Part A: BGB324 400/100 mg: Participants received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 (21 days) followed by a maximum daily maintenance dose of 100 mg thereafter.
- Part A: BGB324 600/200 mg: Participants received daily loading dose of bemcentinib 600 mg on Days 1, 2 and 3 of Cycle 1 (21 days) followed by a maximum daily maintenance dose of 200 mg thereafter.
- Part A: BGB324 900/300 mg: Participants received daily loading dose of bemcentinib 900 mg on Days 1, 2 and 3 of Cycle 1 (21 days) followed by a maximum daily maintenance dose of 300 mg thereafter.
- Part A: BGB324 200/100 mg: Participants received daily loading dose of bemcentinib 200 mg on Days 1, 2 and 3 of Cycle 1 (21 days) followed by a maximum daily maintenance dose of 100 mg thereafter.
- Part A: BGB324 400/200 mg: Participants with AML, received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 (21 days) followed by a maximum daily maintenance dose of 200 mg thereafter.
- B1: BGB324 400/200 mg; B2: BGB324 400/200 mg + Cytarabine: Participants with AML, received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 (21 days) followed by a maximum daily maintenance dose of 200 mg thereafter. In combination to this, participants received cytarabine subcutaneously according to standard practice (20 mg/m^2 twice daily for 10 days followed by a rest period of <1 month according to persisting myelosuppression).
- B3: BGB324 400/200 mg + Decitabine: Participants with AML, received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 (21 days) followed by a maximum daily maintenance dose of 200 mg thereafter. In combination to this, participants received decitabine (up to a maximum dose of 20 mg/m2 body surface area by intravenous infusion over one hour, repeated daily for five consecutive days [i.e., a total of five doses per treatment cycle]).
- B4: BGB324 400/200 mg: Participants with intermediate (int-2) or high risk MDS received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 (21 days) followed by a maximum daily maintenance dose of 200 mg thereafter.
- B5: BGB324 400/200 mg + Cytarabine: Participants with AML, received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 (21 days) followed by a maximum daily maintenance dose of 200 mg thereafter. In combination to this, participants received low dose cytarabine subcutaneously according to standard practice (dose of 20 mg subcutaneously twice daily for 10 days every 28 days).
Arm/Group | Part A: BGB324 400/100 mg | Part A: BGB324 600/200 mg | Part A: BGB324 900/300 mg | Part A: BGB324 200/100 mg | Part A: BGB324 400/200 mg | B1: BGB324 400/200 mg | B2: BGB324 400/200 mg + Cytarabine | B3: BGB324 400/200 mg + Decitabine | B4: BGB324 400/200 mg | B5: BGB324 400/200 mg + Cytarabine
All-Cause Mortality (participants affected / at risk) | 4/6 | 5/14 | 1/5 | 2/4 | 6/7 | 10/14 | 12/16 | 12/18 | 13/18 | 14/20
Serious Adverse Events (participants affected / at risk) | 4/6 | 11/14 | 4/5 | 4/4 | 7/7 | 8/14 | 12/16 | 14/18 | 13/18 | 16/20
Other Adverse Events (participants affected / at risk) | 5/6 | 14/14 | 5/5 | 4/4 | 7/7 | 14/14 | 16/16 | 17/18 | 18/18 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: BGB324 400/100 mg (N=6) | Part A: BGB324 600/200 mg (N=14) | Part A: BGB324 900/300 mg (N=5) | Part A: BGB324 200/100 mg (N=4) | Part A: BGB324 400/200 mg (N=7) | B1: BGB324 400/200 mg (N=14) | B2: BGB324 400/200 mg + Cytarabine (N=16) | B3: BGB324 400/200 mg + Decitabine (N=18) | B4: BGB324 400/200 mg (N=18) | B5: BGB324 400/200 mg + Cytarabine (N=20)
Pneumonia (Infections and infestations) | 2 | 3 | 0 | 1 | 3 | 1 | 1 | 1 | 0 | 3
Lung infection (Infections and infestations) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 2
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary mycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scrotal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 4 | 4 | 5 | 6 | 1 | 5
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral bacterial infection (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial haemorrhage (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1
Glomerulonephritis acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Blood culture positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uncoded (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: BGB324 400/100 mg (N=6) | Part A: BGB324 600/200 mg (N=14) | Part A: BGB324 900/300 mg (N=5) | Part A: BGB324 200/100 mg (N=4) | Part A: BGB324 400/200 mg (N=7) | B1: BGB324 400/200 mg (N=14) | B2: BGB324 400/200 mg + Cytarabine (N=16) | B3: BGB324 400/200 mg + Decitabine (N=18) | B4: BGB324 400/200 mg (N=18) | B5: BGB324 400/200 mg + Cytarabine (N=20)
Diarrhoea (Gastrointestinal disorders) | 1 | 6 | 2 | 2 | 6 | 6 | 6 | 7 | 6 | 11
Nausea (Gastrointestinal disorders) | 3 | 4 | 1 | 1 | 2 | 1 | 4 | 3 | 4 | 11
Vomiting (Gastrointestinal disorders) | 0 | 4 | 3 | 1 | 0 | 3 | 2 | 0 | 2 | 6
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 4
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 2 | 4 | 5 | 0 | 5
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival hyperplasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 1 | 1 | 3
Tongue discolouration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral herpes (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth development disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 2 | 0 | 5 | 2 | 4 | 3 | 1 | 1
Pyrexia (General disorders) | 3 | 7 | 0 | 0 | 2 | 2 | 4 | 3 | 1 | 6
Oedema peripheral (General disorders) | 2 | 2 | 1 | 2 | 0 | 2 | 4 | 3 | 4 | 6
General physical health deterioration (General disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 2
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Night sweats (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Terminal state (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased activity (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 1 | 3 | 2 | 2 | 6 | 6 | 10 | 5 | 10
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 4 | 3 | 1
Weight decreased (Investigations) | 1 | 1 | 1 | 0 | 1 | 0 | 4 | 3 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 1 | 0 | 1 | 2 | 4 | 0 | 1 | 7
White blood cell count increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinomyces test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood chloride increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urine leukocyte esterase positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine increased (Investigations) | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Crystal urine (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fungal test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nitrite urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Red blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scan myocardial perfusion abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 3 | 1 | 5 | 4 | 3 | 5
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 7 | 3 | 3 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymph node calcification (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 6 | 0 | 2 | 1 | 3 | 2 | 4 | 4 | 6
Decreased appetite (Metabolism and nutrition disorders) | 1 | 5 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Iron overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 1 | 2 | 1 | 1 | 4 | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 0 | 0 | 3 | 4 | 2 | 3 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 3 | 2 | 2 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 3 | 2 | 3 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 3
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scrotal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 1 | 0 | 4 | 4 | 0 | 2
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemarthrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 1 | 1 | 3 | 0 | 3 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 3 | 1 | 1 | 2
Dysgeusia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Somnolence (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Orthostatic intolerance (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Movement disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nuchal rigidity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 2 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin wound (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Growing pains (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertonia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Haematoma (Vascular disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 5
Epistaxis (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Skin ulcer (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Intra-abdominal haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tongue haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Venous haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oedema peripheral (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erectile dysfunction (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Food aversion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Amaurosis fugax (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intraocular haematoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scleral haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Penile oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Penile haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulval abscess (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic congestion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Inappropriate antidiuretic hormone secretion (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Anuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urge incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site phlebitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombosis in device (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT02488408/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT02488408/SAP_001.pdf